CLINICAL TRIAL: NCT02994173
Title: Dose Response Study of Patient Controlled Analgesia (PCA) of S-ketamine in Orthopaedic Spine Surgery Patients
Brief Title: Dose-response of Ketamine in Patient Controlled Analgesia in Orthopaedic Surgery Patients
Acronym: DoseRespKeta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T281/2016
Record Dates: First submitted 2016-11-03; First posted 2016-12-15 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Active Comparator): Oxycodone 1 mg / ml alone
  Interventions: Drug: Oxycodone
- Ketamine 0.25 (Active Comparator): Oxycodone 1 mg / ml + S-ketamine 0.25 mg / ml (ratio 1:0.25)
  Interventions: Drug: S-Ketamine 0.25
- Ketamine 0.5 (Active Comparator): Oxycodone 1 mg / ml + S-ketamine 0.5 mg / ml (ratio 1:0.5)
  Interventions: Drug: S-Ketamine 0.5
- Ketamine 0.75 (Active Comparator): Oxycodone 1 mg / ml + S-ketamine 0.75 mg / ml (ratio 1:0.75)
  Interventions: Drug: S-Ketamine 0.75

INTERVENTIONS:
Drug: Oxycodone — Current clinical practice, used as a control in this study
  Other Names: Oxanest
  Arms: Placebo
Drug: S-Ketamine 0.25 — dosage
  Other Names: Ketanest-S
  Arms: Ketamine 0.25
Drug: S-Ketamine 0.5 — dosage
  Other Names: Ketanest-S
  Arms: Ketamine 0.5
Drug: S-Ketamine 0.75 — dosage
  Other Names: Ketanest-S
  Arms: Ketamine 0.75

SUMMARY:
To study the multimodal protocol combining adjunct ketamine with oxycodone in intravenous patient-controlled analgesia bolus dosing and effects in patients scheduled for posterolateral lumbar spine fusion with bilateral transpedicular screw instrumentation

ELIGIBILITY:
Inclusion Criteria:

* 20 - 75 years of age
* Scheduled for elective posterolateral lumbar spine fusion with bilateral transpedicular screw instrumentation under general anaesthesia.
* Written informed consent from the participating patient

Exclusion Criteria:

* A previous history of intolerance to the study drug or related compounds and additives
* Concomitant drug therapy with opioids or strong CYP3A4 or CYP2B6 inductor(s) or inhibitor(s) 2 weeks prior to study.
* Patients younger than 20 years and older than 75 years.
* BMI > 35, sleep apnoea, any other sleep disorder or condition that requires treatment with continuous positive airway pressure or automatic positive airway pressure device.
* Existing significant liver or kidney disease
* History of ischemic heart disease or conduction disturbance
* History of alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent
* Donation of blood for 4 weeks prior and during the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change in opioid consumption (mg) postoperatively | 24 and 72 hours
  Change from baseline opioid consumption (mg) postoperatively at 24 and 72 hours

SECONDARY OUTCOMES:
Change in numerical rating scale (NRS 0-10) | 24 and 72 hours
  Change from baseline NRS value postoperatively at 24 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marko Peltoniemi, MD, PhD, Principal Investigator — Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital
Locations (1):
- Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No